CLINICAL TRIAL: NCT00458848
Title: Phase II Study of Adult Acute Lymphoblastic Leukaemia (ALL): Imatinib in Combination With Chemotherapy in Ph+ Patients, and Post-remissional Treatment Intensification in High-risk Ph- Patients, With Minimal Residual Disease Monitoring.
Brief Title: Chemotherapy With or Without Imatinib and/or Peripheral Stem Cell Transplant in Acute Lymphoblastic Leukemia
Acronym: LAL0904
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL0904; LAL0904 (Other: GIMEMA); 2004-001738-11 (Other: EudraCT)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Leukemia
Keywords: B-cell adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; TdT positive adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Daunorubicin; Etoposide; Idarubicin; Imatinib Mesylate; Mercaptopurine; Methotrexate; Methylprednisolone; Mitoxantrone; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: asparaginase
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: idarubicin
Drug: imatinib mesylate
Drug: mercaptopurine
Drug: methotrexate
Drug: methylprednisolone
Drug: mitoxantrone hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: autologous hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. When the healthy stem cells are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving combination chemotherapy together with imatinib mesylate and peripheral stem cell transplant may be an effective treatment for acute lymphoblastic leukemia.

Nevertheless, in the last few years GIMEMA has pubblished a paper in which 100% of Ph+ ALL patients reach HCR only with Imatinib, without any chemiotherapy. Thus, this treatment will be implemented in patients pertaining to this category.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL) meeting the following criteria:

  * Negative myeloperoxidase stain
  * Phenotype T (T-ALL) or B (B-ALL)
  * No mature B-ALL (FAB L3, serum immunoglobulin-positive, terminal deoxynucleotidyl transferase-negative)

PATIENT CHARACTERISTICS:

* Creatinine ≤ 2.5 mg/dL (after adequate hydration)
* SGOT and SGPT ≤ 3 times upper limit of normal
* LVEF ≥ 50%
* No severe psychiatric disorders
* No other concurrent malignant disease
* No presence of documented infections not responding to antibiotic and/or antifungal therapy
* Not pregnant

PRIOR CONCURRENT THERAPY:

* No prior steroids
* No prior antiblastic chemotherapy
* No other concurrent chemotherapy or radiotherapy

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 470 (Actual)
Dates: Start 2004-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foa, MD, Study Chair — Universita Degli Studi "La Sapeinza"
Locations (66):
- Italy (66):
  - Ospedale Civile Alessandria, Alessandria
  - Ospedale Torrette University Ancona, Ancona
  - Ospedale S. Donato, Arezzo
  - Dipartimento Area Medica - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - S.G. Moscati Hospital, Avellino
  - Universita Degli Studi di Bari, Bari
  - University of Bologna Medical School, Bologna
  - Spedali Civili di Brescia, Brescia
  - A. Perrino Hospital, Brindisi
  - Ospedale Binaghi, Cagliari
  - Ospedale Ferrarotto, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - Universita di Ferrara, Ferrara
  - Azienda Ospedaliera di Firenze, Florence
  - Ospedali Riuniti Foggia, Foggia
  - Ospedale Umberto I, Frosinone
  - Ospedale S. Antonio Abate, Gallarate
  - Ospedale San Martino, Genoa
  - Ospedale Santa Maria Goretti, Latina
  - Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Ospedale Maggiore Lodi, Lodi
  - Ospedale L'Aquila, L’Aquila
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino, Messina
  - Ospedale Niguarda Ca'Granda, Milan
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - Azienda Ospedaliera di Rilievo Nazionale A.Cardarelli, Naples
  - Federico II University Medical School, Naples
  - Ospedale S. Gennaro ASL NA1, Naples
  - Inferiore U.O. Medicina Interna Ematologia ed Oncologia P.O. Umberto I, Nocera Inferiore
  - Amedeo Avogadro University of Eastern Piedmont, Novara
  - Ospedale San Francesco, Nuoro
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico - Cattedra di Ematologia, Palermo
  - Ospedale Cervello, Palermo
  - Ospedale La Maddalena - Palermo, Palermo
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - University of Pavia, Pavia
  - Perugia Regional Cancer Center, Perugia
  - Azienda Ospedale - d S. Salvatore, Pesaro
  - Ospedale Civile Pescara, Pescara
  - Azienda Ospedaliera Pisana, Pisa
  - Azienda Ospedaliera San Carlo - Potenza, Potenza
  - Ospedale Sta. Maria Delle Croci, Ravenna
  - Ospedale S. M. delle Croci, Ravenna
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale Oncologico Regionale, Rionero in Vulture
  - Ospedale Sant' Eugenio, Rome
  - Azienda Ospedaliera S. Camillo-Forlanini, Rome
  - University Campus Bio-Medico, Rome
  - Istituto Regina Elena, Rome
  - Universita Degli Studi "La Sapeinza", Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - H. San Giovanni-Addolorata Hospital, Rome
  - Ospedale di Ronciglione, Ronciglione
  - IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - Istituto di Ematologia Universita - University di Sassari, Sassari
  - Azienda Ospedale E. Morelli, Sondalo
  - Ospedale S. Vincenzo, Taormina
  - Ospedal SS Annunziata, Taranto
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
  - Ospedale Giovanni Bosco, Turin
  - Policlinico Universitario Udine, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

REFERENCES:
- [Background] Chiaretti S, Vitale A, Vignetti M, Piciocchi A, Fazi P, Elia L, Falini B, Ronco F, Ferrara F, De Fabritiis P, Luppi M, La Nasa G, Tedeschi A, Califano C, Fanin R, Dore F, Mandelli F, Meloni G, Foa R. A sequential approach with imatinib, chemotherapy and transplant for adult Ph+ acute lymphoblastic leukemia: final results of the GIMEMA LAL 0904 study. Haematologica. 2016 Dec;101(12):1544-1552. doi: 10.3324/haematol.2016.144535. Epub 2016 Aug 11. PMID 27515250
- [Result] Messina M, Chiaretti S, Iacobucci I, Tavolaro S, Lonetti A, Santangelo S, Elia L, Papayannidis C, Paoloni F, Vitale A, Guarini A, Martinelli G, Foa R. AICDA expression in BCR/ABL1-positive acute lymphoblastic leukaemia is associated with a peculiar gene expression profile. Br J Haematol. 2011 Mar;152(6):727-32. doi: 10.1111/j.1365-2141.2010.08449.x. Epub 2011 Jan 31. PMID 21623761
- [Derived] Piciocchi A, Messina M, Elia L, Vitale A, Soddu S, Testi AM, Chiaretti S, Mancini M, Albano F, Spadano A, Krampera M, Bonifacio M, Cairoli R, Vetro C, Colella F, Ferrara F, Cimino G, Bassan R, Fazi P, Vignetti M. Prognostic impact of KMT2A-AFF1-positivity in 926 BCR-ABL1-negative B-lineage acute lymphoblastic leukemia patients treated in GIMEMA clinical trials since 1996. Am J Hematol. 2021 Sep 1;96(9):E334-E338. doi: 10.1002/ajh.26253. Epub 2021 Jun 9. No abstract available. PMID 34048072
- See also: GIMEMA Foundation Website — http://www.gimema.it

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We are reporting on the subset of patients that was treated according to amendment three, in which Imatinib was given only at induction.
Groups:
- Philadelphia Positive, Imatinib Only in Induction Therapy: These subset of patients was treated according to amendment three, in which Imatinib was given only at induction.
Period: Overall Study
Arm/Group | Philadelphia Positive, Imatinib Only in Induction Therapy
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Philadelphia Positive, Imatinib Only in Induction Therapy: In this protocol, adult Philadelphia positive acute lymphoblastic leukemia patients were treated with chemotherapy for induction and consolidation, followed by maintenance with imatinib. The protocol was subsequently amended and imatinib was incorporated in the induction and post-remission phase together with chemotherapy. Due to the toxicity of this combined approach, the protocol was further amended to a sequential scheme based on imatinib plus steroids as induction, followed by consolidation with chemotherapy plus imatinib and, when applicable, by a hematopoietic stem cell transplant.
  Thus, we have analyzed only this subset of patients as it was not feasible to analyzed all patients enrolled due also to the disease itself.
Arm/Group | Philadelphia Positive, Imatinib Only in Induction Therapy
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 45.94 [16.99 to 59.70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 51
White Blood Cells (WBC) at diagnosis-nsr [Median (Full Range); unit: 10^9 cells/L] | 28.00 [1.40 to 597.00]
BCR transcript-molecular at diagnosis [Number; unit: participants]
  p190 | 39
  p210 | 7
  p190/p210 | 5
Pre-treatment response [Number; unit: participants]
  Non responder-blasts reduction <75% | 10
  Responder-blasts reduction >=75% | 38
  Frequency missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reaching Disease Free Survival
Time Frame: At 60 months
Measure: Number; unit: percentage of participants
Arm/Group | Philadelphia Positive, Imatinib Only in Induction Therapy
Number analyzed (Participants) | 51
percentage of participants | 45.8

2. Secondary Outcome: Number of Patients Reaching Complete Hematological Response After Induction Therapy
Time Frame: At the end of induction, day +50
Measure: Number; unit: participants
Arm/Group | Philadelphia Positive, Imatinib Only in Induction Therapy
Number analyzed (Participants) | 51
participants | 49

3. Secondary Outcome: Percentage of Participants Reaching Overall Survival
Description: Overall survival from diagnosis
Time Frame: At 60 months
Measure: Number; unit: percentage of patients
Arm/Group | Philadelphia Positive, Imatinib Only in Induction Therapy
Number analyzed (Participants) | 51
percentage of patients | 48.8

ADVERSE EVENTS:
Time Frame: 34 months
Description: Only serious adverse events are reported.
Arm/Group | Philadelphia Positive, Imatinib Only in Induction Therapy
All-Cause Mortality (participants affected / at risk) | 2/51
Serious Adverse Events (participants affected / at risk) | 7/51
Other Adverse Events (participants affected / at risk) | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Philadelphia Positive, Imatinib Only in Induction Therapy (N=51)
Death (General disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No